CLINICAL TRIAL: NCT01004250
Title: A Single-Arm, Phase 2 Trial of Pemetrexed, Cisplatin,and Bevacizumab as Induction, Followed by Pemetrexed and Bevacizumab as Maintenance, in First-Line Treatment of Nonsquamous Advanced NSCLC
Brief Title: A Study of Pemetrexed and Bevacizumab for Participants With Advanced Non-Small Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13034; H3E-EW-S125 (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Treatment (Experimental)
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Pemetrexed — 500 milligram per square meter (mg/m²) given intravenously on Day 1 of each 21-day cycle for four cycles of Induction Therapy, and continued in Maintenance Therapy until progression or unacceptable toxicity.
  Other Names: Alimta; LY231514
Drug: Cisplatin — 75 mg/m² given intravenously on Day 1 of 21-day cycle for a maximum of 4 cycles
Drug: Bevacizumab — 7.5 milligram per kilogram (mg/kg) given intravenously on Day 1 of 21-day cycle for four cycles of Induction Therapy, and continued in Maintenance Therapy until progression or unacceptable toxicity

SUMMARY:
Participants with advanced non-small cell lung cancer (NSCLC) will receive a first-line treatment of Pemetrexed, Cisplatin and Bevacizumab as induction therapy followed by a maintenance treatment of Pemetrexed and Bevacizumab. Treatment will continue until disease progression or unacceptable toxicity occurs. The primary objective of this study is to measure how long this treatment could prevent the disease progression.

DETAILED DESCRIPTION:
The study will have 3 periods: a baseline period; a study treatment period, including both induction and maintenance treatment; and a follow-up period. Approximately 110 participants will be enrolled into the study, with the aim of having 100 evaluable participants. Eligible participants will first receive 4 cycles of induction chemotherapy with pemetrexed-cisplatin-bevacizumab. Participants who achieve a response or do not progress after completion of induction chemotherapy and have an adequate performance status will receive maintenance therapy with pemetrexed-bevacizumab. Treatment will continue until disease progression or unacceptable toxicity occurs. When treatment is discontinued, the participants health status will be monitored till death, loss to follow-up or data cut-off date.

Participants who continue to receive benefit from treatment at the time of data cut-off may receive continued access to pemetrexed and bevacizumab until disease progression, unacceptable toxicity, or any other reason at investigator or participants decision.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of nonsquamous Stage IIIB or Stage IV NSCLC that is not amenable to curative therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* At least 1 unidimensionally measurable lesion meeting the Response Evaluation Criteria In Solid Tumors (RECIST) criteria
* Adequate organ function, including the following:

  * Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) ≥1.5 x 10^9 per Liter (10^9/L), platelets ≥100 x 10^9/L, and hemoglobin ≥10 gram per deciliter (g/dL)
  * Hepatic: bilirubin ≤1.5 times the upper limit of normal (ULN); alkaline phosphatase (AP), aspartate aminotransferase (AST), and alanine aminotransferase (ALT) ≤3.0 x ULN (AP, AST, and ALT ≤5 x ULN is acceptable if liver has tumor involvement)
  * Renal: calculated creatinine clearance (CrCl) ≥45 milliliter per minute (mL/min) based on the original weight-based Cockcroft and Gault formula, and serum creatinine ≤1.5 x ULN
  * At the time of enrollment, if the urinalysis dipstick result is ≥2+ for protein, a 24-hour urine collection should be taken. In these cases, participants must have ≤1g protein/24 hours to be eligible for study participation
* Participants must sign an Informed Consent Document (ICD)

Exclusion Criteria:

* Have received prior systemic anticancer therapy for lung cancer (including adjuvant early-stage treatment for NSCLC)
* Have a serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease, as defined by the New York Heart Association Class III or IV
* Have a second primary malignancy that is clinically detectable at the time of consideration for study enrollment
* Have known central nervous system (CNS) disease, other than stable, treated brain metastasis. Stable, treated brain metastasis is defined as metastasis having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and post-treatment brain imaging (Computed Tomography [CT] scan or magnetic resonance imaging [MRI])
* Are receiving concurrent administration of any other antitumor therapy
* Have a history of gastrointestinal fistula, perforation, or abscess, inflammatory bowel disease, or diverticulitis
* Have had significant weight loss (that is, ≥10%) over the previous 6 weeks before study entry
* Have a history of gross hemoptysis (bright red blood of ≥½ teaspoon per episode of coughing) <3 months prior to enrollment or history or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding
* Are taking or have recently taken (within 10 days of enrollment) full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes. Prophylactic use of anticoagulants is allowed; international normalized ratio (INR) should be <1.5 at study enrollment
* Have a history of hypertension, unless hypertension is well controlled upon study entry (≤150/90 millimeter of mercury [mm Hg]) and the participant is on a stable regimen of antihypertensive therapy. Participants should not have any prior history of hypertensive crisis or hypertensive encephalopathy
* Have had major surgery, open biopsy, or significant traumatic injury within 28 days prior to study enrollment, or anticipate the need for major surgical procedure during the course of the study
* History of thrombotic disorders within the last 6 months prior to entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2009-10; Primary Completion 2012-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (19):
- Denmark (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Copenhagen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herlev
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coswig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Magdeburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lecce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rozzano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trento
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaén
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pozuelo de Alarcón
- Sweden (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Solna

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had 3 periods: a baseline period; a study treatment period, including both induction (Ind) and maintenance (Maint) treatment; and a follow-up period.
Groups:
- Study Treatment: Induction Therapy:
  Bevacizumab: 7.5 milligram per kilogram (mg/kg) given intravenously on Day 1 for four cycles (cycle=21 days) of Induction Therapy.
  Pemetrexed: 500 milligram per square meter (mg/m²) given intravenously on Day 1 for four cycles of Induction Therapy.
  Cisplatin: 75 mg/m² given intravenously on Day 1 for a maximum of 4 cycles.
  Maintenance Therapy:
  Bevacizumab: 7.5 mg/kg given intravenously on Day 1 of each cycle (cycle=21 days) and continued until progression or unacceptable toxicity.
  Pemetrexed: 500 mg/m² given intravenously on Day 1 of each cycle and continued until progression or unacceptable toxicity.
Period: Induction Therapy Period
Arm/Group | Study Treatment
Started | 109
Received at Least One Dose of Study Drug | 109
Death (Any Cause) or Disease Progression | 21 (Participants (pts) with death or disease progression considered to have completed phase.)
Completed | 94
Not Completed | 15
Not completed — Adverse Event | 10
Not completed — Entry Criteria Not Met | 1
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2
Period: Maintenance Therapy Period
Arm/Group | Study Treatment
Started | 72 (Did not enter Maint: 21 pts due to death or disease progression; 1 pts had performance status 2.)
Death (Any Cause) or Disease Progression | 46 (Pts with death or disease progression considered to have completed phase.)
Completed | 46
Not Completed | 26
Not completed — Adverse Event | 15
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 4
Period: Follow-Up (FU) Period
Arm/Group | Study Treatment
Started | 101 (Did not enter FU:Death-4pts Ind,1pts Maint; Pt Withdrew-1 pts Ind,1pts Maint; Lost to FU-1 pts Maint)
Completed | 100
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Intent To Treat population who receive at least 1 dose of study drug.
Groups:
- Study Treatment: Induction Therapy:
  Bevacizumab: 7.5 mg/kg given intravenously on Day 1 for four cycles (cycle=21 days) of Induction Therapy.
  Pemetrexed: 500 mg/m² given intravenously on Day 1 for four cycles of Induction Therapy.
  Cisplatin: 75 mg/m² given intravenously on Day 1 for a maximum of 4 cycles.
  Maintenance Therapy:
  Bevacizumab: 7.5 mg/kg given intravenously on Day 1 of each cycle and continued until progression or unacceptable toxicity.
  Pemetrexed: 500 mg/m² given intravenously on Day 1 of each cycle and continued until progression or unacceptable toxicity.
Arm/Group | Study Treatment
Number analyzed (Participants) | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 108
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 12
  Denmark | 19
  Germany | 25
  Italy | 35
  Sweden | 18
ECOG Performance Status [Number; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status Classifies participants according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death):
  0 - Fully Active
  1. - Ambulatory, Restricted Strenuous Activity
  2. - Ambulatory, No Work Activities
  3. - Partially Confined to Bed, Limited Self Care
  4. - Completely Disabled
  5. - Death
  Participants
    ECOG 0 | 59
    ECOG 1 | 50
Initial Pathological Diagnosis [Number; unit: Participants] — Non-Small Cell Lung Cancer (NSCLC)
  Participants
    Adenocarcinoma | 99
    Large Cell Lung Carcinoma | 3
    Poorly Differentiated NSCLC | 3
    Other | 4
Stage of Disease [Number; unit: Participants] — According to American Joint Committee on Cancer (AJCC) Cancer Staging Manual, sixth edition (2002), stage of disease means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body).
  Stage IIIB - the cancer has spread to nearby tissue or spread to far away lymph nodes but not spread to other organs
  Stage IV - the cancer has spread to other organs of the body such as the other lung, brain, or liver
  Participants
    Stage IIIB | 10
    Stage IV | 99
Tobacco Use [Number; unit: Participant]
  Never Smoked | 15
  Ex-Smoker | 66
  Current Smoker | 28

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression-Free Survival (PFS) is defined as the time from the date of study enrollment to the first date of objectively determined PD or death from any cause. PD is defined using Response Evaluation Criteria in Solid Tumours (RECIST) Guidelines (Version 1.0), as at least a 20% increase in the sum of longest diameter (LD) of target lesions, taking as references the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions. For participants not known to have died as of the data cut-off date and who do not have objective PD, PFS will be censored at the date of the last objective progression-free disease assessment. For participants who receive subsequent systemic anticancer therapy, PFS will be censored at the date of the last objective progression-free disease assessment prior to post-discontinuation systemic therapy.
Time Frame: From enrollment to the first date of objectively determined Progressive Disease (PD) or death from any cause (every other cycle during study treatment and then every 6 weeks during follow-up period)(Baseline up to 36.1 Months)
Population: 30 participants were censored. Participants qualified by the following criteria:
  * Confirmed histological or cytological diagnosis of nonsquamous Stage IIIB or Stage IV lung cancer
  * At least 1 unidimensionally measurable lesion
  * No concomitant curative anticancer therapy
  * Treated with at least one dose of study drug
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Study Treatment
Number analyzed (Participants) | 109
Months | 6.9 [5.7 to 8.3]

2. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from the date of study enrollment to the date of death from any cause. For participants not known to have died as of the data cut-off date, OS will be censored at the last contact date.
Time Frame: From enrollment to the date of death from any cause (every cycle during study treatment, every 6 weeks during follow-up period until PD, and then at least every 3 Months) (Baseline up to 36.3 Months)
Population: 32 participants were censored. All enrolled participants receiving at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Study Treatment
Number analyzed (Participants) | 109
Months | 14.7 [11.5 to 19.7]

3. Secondary Outcome: Percentage of Participants With Confirmed Complete Response or Partial Response During Study Treatment (Induction and Maintenance)
Description: Overall Response Rate (ORR) is defined as the percentage of participants whose best response is complete response (CR) or partial response (PR) per RECIST Guidelines, Version 1.0. CR is disappearance of all tumor lesions. PR is either a) at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LDs, or b) complete disappearance of target lesions, with persistence (but not worsening) of 1 or more nontarget lesions. In either case, no new lesions may have appeared.
Time Frame: From enrollment to objectively determined PD (assessment during study treatment completed at every other cycle till PD and at 30 day follow-up)(Baseline up to 104.1 Weeks)
Population: Participants qualified by the following criteria:
  * Confirmed histological or cytological diagnosis of nonsquamous Stage IIIB or Stage IV lung cancer
  * At least 1 unidimensionally measurable lesion
  * No concomitant curative anticancer therapy
  * Treated with at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Study Treatment
Number analyzed (Participants) | 109
Percentage of Participants | 42.2 [32.8 to 52.0]

4. Secondary Outcome: Percentage of Participants With Confirmed Response Complete or Partial Response During the Induction Treatment Only
Description: CR and PR defined per RECIST Guidelines, Version 1.0. CR is disappearance of all tumor lesions. PR is either a) at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LDs, or b) complete disappearance of target lesions, with persistence (but not worsening) of 1 or more nontarget lesions. In either case, no new lesions may have appeared.
Time Frame: From the time of study enrollment to the first date of objectively determined PD during the induction therapy (assessment during study treatment completed at every other cycle up to four cycles) (Baseline up to 4 cycles)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Study Treatment: Induction Therapy:
  Bevacizumab: 7.5 mg/kg given intravenously on Day 1 for four cycles (cycle=21 days) of Induction Therapy.
  Pemetrexed: 500 mg/m² given intravenously on Day 1 for four cycles of Induction Therapy.
  Cisplatin: 75 mg/m² given intravenously on Day 1 for a maximum of 4 cycles.
Arm/Group | Study Treatment
Number analyzed (Participants) | 109
Percentage of Participants | 34.9 [26.0 to 44.6]

5. Secondary Outcome: Percentage of Participants With Confirmed Complete Response or Partial Response During the Maintenance Therapy Only
Description: as for outcome 4
Time Frame: From the start of the maintenance to the first date of objectively determined PD during the maintenance therapy (assessment during maintenance treatment completed at every other cycle till PD and at 30 day follow-up)(Cycle 5 up to 104.1 Weeks)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Study Treament: Induction Therapy:
  Bevacizumab: 7.5 mg/kg given intravenously on Day 1 for four cycles (cycle=21 days) of Induction Therapy.
  Pemetrexed: 500 mg/m² given intravenously on Day 1 for four cycles of Induction Therapy.
  Cisplatin: 75 mg/m² given intravenously on Day 1 for a maximum of 4 cycles.
  Maintenance Therapy:
  Bevacizumab: 7.5 mg/kg given intravenously on Day 1 of each cycle and continued until progression or unacceptable toxicity.
  Pemetrexed: 500 mg/m² given intravenously on Day 1 of each cycle and continued until progression or unacceptable toxicity.
Arm/Group | Study Treament
Number analyzed (Participants) | 72
Percentage of Participants | 11.1 [4.9 to 20.7]

ADVERSE EVENTS:
Groups:
- Induction Therapy: Induction Therapy:
  Bevacizumab: 7.5 mg/kg given intravenously on Day 1 for four cycles (cycle=21 days) of Induction Therapy.
  Pemetrexed: 500 mg/m² given intravenously on Day 1 for four cycles of Induction Therapy.
  Cisplatin: 75 mg/m² given intravenously on Day 1 for a maximum of 4 cycles.
- Maintenance Therapy: Maintenance Therapy:
  Bevacizumab: 7.5 mg/kg given intravenously on Day 1 of each cycle and continued until progression or unacceptable toxicity.
  Pemetrexed: 500 mg/m² given intravenously on Day 1 of each cycle and continued until progression or unacceptable toxicity.
- Overall Study Treatment: Induction Therapy:
  Bevacizumab: 7.5 mg/kg given intravenously on Day 1 for four cycles (cycle=21 days) of Induction Therapy.
  Pemetrexed: 500 mg/m² given intravenously on Day 1 for four cycles of Induction Therapy.
  Cisplatin: 75 mg/m² given intravenously on Day 1 for a maximum of 4 cycles.
  Maintenance Therapy:
  Bevacizumab: 7.5 mg/kg given intravenously on Day 1 of each cycle and continued until progression or unacceptable toxicity.
  Pemetrexed: 500 mg/m² given intravenously on Day 1 of each cycle and continued until progression or unacceptable toxicity.
Arm/Group | Induction Therapy | Maintenance Therapy | Overall Study Treatment
Serious Adverse Events (participants affected / at risk) | 32/109 | 14/72 | 39/109
Other Adverse Events (participants affected / at risk) | 105/109 | 68/72 | 106/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Therapy (N=109) | Maintenance Therapy (N=72) | Overall Study Treatment (N=109)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) — Event resulted in death
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Asthenia (General disorders) | 1 (1) | 1 (1) | 2 (2)
Chest pain (General disorders) | 2 (2) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 4 (4) | 1 (1) | 5 (5)
Sudden death (General disorders) | 1 (1) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) — Event resulted in 1 death
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Therapy (N=109) | Maintenance Therapy (N=72) | Overall Study Treatment (N=109)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 1 (1) | 9 (9)
Leukopenia (Blood and lymphatic system disorders) | 9 (15) | 4 (12) | 11 (31)
Neutropenia (Blood and lymphatic system disorders) | 18 (29) | 12 (27) | 22 (60)
Palpitations (Cardiac disorders) | 0 (0) | 4 (4) | 4 (4)
Tinnitus (Ear and labyrinth disorders) | 9 (10) | 2 (2) | 11 (12)
Lacrimation increased (Eye disorders) | 11 (11) | 7 (9) | 16 (19)
Constipation (Gastrointestinal disorders) | 28 (33) | 16 (21) | 39 (54)
Diarrhoea (Gastrointestinal disorders) | 17 (18) | 11 (12) | 25 (29)
Dyspepsia (Gastrointestinal disorders) | 9 (10) | 6 (6) | 14 (15)
Gastritis (Gastrointestinal disorders) | 3 (3) | 4 (4) | 6 (7)
Nausea (Gastrointestinal disorders) | 60 (100) | 17 (27) | 64 (128)
Stomatitis (Gastrointestinal disorders) | 9 (13) | 9 (12) | 17 (25)
Vomiting (Gastrointestinal disorders) | 21 (28) | 10 (17) | 25 (45)
Asthenia (General disorders) | 5 (6) | 4 (6) | 9 (12)
Chest pain (General disorders) | 7 (7) | 3 (3) | 9 (10)
Fatigue (General disorders) | 42 (47) | 20 (22) | 51 (63)
Influenza like illness (General disorders) | 1 (1) | 6 (6) | 7 (7)
Mucosal inflammation (General disorders) | 12 (15) | 5 (6) | 14 (20)
Oedema peripheral (General disorders) | 5 (5) | 10 (10) | 14 (14)
Pain (General disorders) | 2 (2) | 5 (5) | 7 (7)
Pyrexia (General disorders) | 11 (12) | 9 (22) | 17 (34)
Infection (Infections and infestations) | 2 (2) | 4 (5) | 6 (7)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (4) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 7 (8) | 8 (10)
Blood creatinine increased (Investigations) | 0 (0) | 7 (7) | 7 (7)
Haemoglobin decreased (Investigations) | 3 (3) | 5 (5) | 7 (9)
Weight decreased (Investigations) | 8 (8) | 4 (4) | 11 (11)
Decreased appetite (Metabolism and nutrition disorders) | 9 (10) | 15 (18) | 22 (29)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 9 (12) | 10 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (8) | 12 (12)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 6 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (7) | 6 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (8) | 7 (9)
Dizziness (Nervous system disorders) | 5 (5) | 5 (5) | 10 (11)
Dysgeusia (Nervous system disorders) | 5 (5) | 5 (5) | 10 (10)
Headache (Nervous system disorders) | 12 (12) | 10 (11) | 19 (22)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 4 (6) | 6 (9)
Paraesthesia (Nervous system disorders) | 7 (7) | 4 (4) | 10 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (9) | 10 (12) | 17 (20)
Anxiety (Psychiatric disorders) | 3 (3) | 3 (3) | 6 (6)
Insomnia (Psychiatric disorders) | 8 (8) | 4 (4) | 12 (12)
Proteinuria (Renal and urinary disorders) | 5 (5) | 3 (4) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 15 (19) | 22 (29)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 15 (19) | 16 (22)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 14 (19) | 28 (38)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (8) | 8 (9)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (2) | 8 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (7) | 11 (16)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 6 (8) | 8 (11)
Hypertension (Vascular disorders) | 14 (14) | 14 (16) | 23 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days